CLINICAL TRIAL: NCT01241240
Title: Safety and Efficacy of Triple Combination Therapy in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-063
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple Combination Therapy (Experimental): Triple Combination Therapy with bimatoprost/brimonidine tartrate/timolol ophthalmic solution. One drop of Triple Combination Therapy administered to each eye, twice daily for 12 weeks.
  Interventions: Drug: bimatoprost/brimonidine tartrate/timolol ophthalmic solution (Triple Combination Therapy)
- Combigan® (Active Comparator): Fixed Combination brimonidine tartrate/timolol ophthalmic solution (Combigan®). One drop of Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution administered to each eye, twice daily for 12 weeks.
  Interventions: Drug: Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost/brimonidine tartrate/timolol ophthalmic solution (Triple Combination Therapy) — One drop of Triple Combination Therapy administered to each eye, twice daily for 12 weeks.
  Arms: Triple Combination Therapy
Drug: Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution — One drop of Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution administered to each eye, twice daily for 12 weeks.
  Other Names: COMBIGAN®
  Arms: Combigan®

SUMMARY:
This study will evaluate the safety and efficacy of Triple Combination Therapy compared with Fixed Combination brimonidine tartrate/timolol ophthalmic solution in patients with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or primary open-angle glaucoma in each eye
* Requires treatment with IOP-lowering medication in both eyes

Exclusion Criteria:

* Required chronic use of ocular medications during the study other than study medication
* Use of any corticosteroids within 30 days
* History of any prior eye surgery, except for uncomplicated eye surgery performed more than 6 months before the Screening visit
* Anticipated wearing of contact lenses during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Bogotá, Colombia
- Mexico City, Mexico

REFERENCES:
- [Derived] Hartleben C, Parra JC, Batoosingh A, Bernstein P, Goodkin M. A Masked, Randomized, Phase 3 Comparison of Triple Fixed-Combination Bimatoprost/Brimonidine/Timolol versus Fixed-Combination Brimonidine/Timolol for Lowering Intraocular Pressure. J Ophthalmol. 2017;2017:4586763. doi: 10.1155/2017/4586763. Epub 2017 Sep 19. PMID 29057117

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triple Combination Therapy | Combigan®
Started | 94 | 98
Completed | 86 | 89
Not Completed | 8 | 9
Not completed — Adverse Event | 5 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Personal Reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple Combination Therapy | Combigan® | Total
Number analyzed (Participants) | 94 | 98 | 192
Age, Customized [Number; unit: Participants]
  ≤65 years | 67 | 74 | 141
  >65 years | 27 | 24 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 73 | 151
  Male | 16 | 25 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Worse Eye Intraocular Pressure (IOP) at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. For each eye, the IOP was either the average of 2 measurements, or, if a third measurement was required, the median of the 3 measurements. The worse eye was determined based on the IOP results at Baseline. The mean worse eye IOP was the average of the IOP measurements of the worse eye at hours 0 and 2 at week 12. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Participants from the modified Intent-to-treat (mITT) population, that included all randomized participants who had at least 1 post-baseline IOP measurement, with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Triple Combination Therapy | Combigan®
Number analyzed (Participants) | 93 | 97
mmHg
  Baseline (n=93,95) | 24.62 (2.475) | 25.12 (2.178)
  Change from Baseline at Week 12 (n=93,94) | -10.03 (2.661) | -9.18 (2.566)

2. Secondary Outcome: Change From Baseline in Mean Worse Eye IOP
Description: IOP is a measurement of the fluid pressure inside the eye. For each eye, the IOP was either the average of 2 measurements, or, if a third measurement was required, the median of the 3 measurements. The worse eye was determined based on the IOP results at Baseline. The mean worse eye IOP was the average of the IOP measurements of the worse eye at hours 0 and 2 at each visit. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 1, 2, 4 and 8
Population: Participants from the mITT population, that included all randomized participants who had at least 1 post-baseline IOP measurement, with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Triple Combination Therapy | Combigan®
Number analyzed (Participants) | 93 | 97
mmHg
  Baseline (n=93,95) | 24.62 (2.475) | 25.12 (2.178)
  Change from Baseline at Week 1 (n=91,89) | -10.18 (3.149) | -8.90 (3.044)
  Change from Baseline at Week 2 (n=88,93) | -10.40 (2.802) | -9.06 (2.925)
  Change from Baseline at Week 4 (n=86,90) | -10.06 (2.793) | -9.21 (2.306)
  Change from Baseline at Week 8 (n=88,89) | -9.77 (2.852) | -9.02 (2.869)

3. Secondary Outcome: Mean Worse Eye IOP
Description: IOP is a measurement of the fluid pressure inside the eye. For each eye, the IOP was either the average of 2 measurements, or, if a third measurement was required, the median of the 3 measurements. The worse eye was determined based on the IOP results at Baseline. The mean worse eye IOP was the average of the IOP measurements of the worse eye at hours 0 and 2 at each time-point.
Time Frame: Weeks 1, 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Triple Combination Therapy | Combigan®
Number analyzed (Participants) | 93 | 97
mmHg
  Week 1 (n=91,90) | 14.43 (2.785) | 16.23 (2.968)
  Week 2 (n=88,95) | 14.05 (2.634) | 16.08 (2.726)
  Week 4 (n=86,92) | 14.38 (2.587) | 15.96 (2.705)
  Week 8 (n=88,91) | 14.68 (2.709) | 16.11 (2.935)
  Week 12 (n=86,88) | 14.43 (2.344) | 15.92 (2.867)

ADVERSE EVENTS:
Description: The Safety Population, all participants who received at least one dose of study drug and had at least one post-baseline visit, was used to assess Serious Adverse Events and Adverse Events.
Arm/Group | Triple Combination Therapy | Combigan®
Serious Adverse Events (participants affected / at risk) | 3/93 | 0/98
Other Adverse Events (participants affected / at risk) | 57/93 | 25/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=93) | Combigan® (N=98)
Bradycardia (Cardiac disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyomyositis (Infections and infestations) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=93) | Combigan® (N=98)
Conjunctival hyperaemia (Eye disorders) | 22 | 4
Eye irritation (Eye disorders) | 13 | 4
Dry eye (Eye disorders) | 10 | 2
Eye pruritus (Eye disorders) | 6 | 2
Somnolence (Nervous system disorders) | 5 | 8
Visual field defect (Nervous system disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release. No documents containing confidential information from the sponsor or information developed will be submitted for publication without prior written authorization from the sponsor.